CLINICAL TRIAL: NCT05500989
Title: PlacEntal Acute Atherosis RefLecting Subclinical Atherosclerosis
Acronym: PEARLS
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Modified NL52556.068.15; METC 152019 (Other: Local Ethical Organisation)
Record Dates: First submitted 2022-05-05; First posted 2022-08-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pre-Eclampsia; HELLP Syndrome; Intrauterine Growth Restriction; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for biomarker analyses
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (6):
- Short track controls: Controls are women (18 years or older) with an uncomplicated pregnancy (i.e no foetal or maternal placental complications, such as pregnancy induced hypertension, preeclampsia or HELLP-syndrome, or small for gestational birth infancies).
  Follow up roughly 18 months postpartum.
- Short track early PE with IUGR: These cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivided into early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Follow up roughly 18 months postpartum.
- Short track early PE without IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivided into early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Follow up roughly 18 months postpartum.
- Short track late PE with IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivided into early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Follow up roughly 18 months postpartum.
- Short track late PE without IUGR: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivided into early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Follow up roughly 18 months postpartum.
- Long term follow up track cases: Cases consist of women (18 years or older) with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (PE is defined as hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with de novo proteinuria (≥ 300 mg/ 24 hours)) Cases will be subdivided into early and late PE, with or without IUGR (Early PE is defined as the occurence of PE < 34 weeks of gestation, whereas late PE is defined as the occurence of PE ≥ 34 weeks of gestation. IUGR is defined as birthweight below the 10th percentile).
  Follow up roughly 18 months postpartum.

SUMMARY:
Pregnancy is considered a cardiovascular (CV) stress test, and complicated pregnancies are associated with an increased risk for cardiovascular disease (CVD) later in life. Moreover, it is known that often the pregnancy induced CV adaptation does not resolve completely after a short postpartum (PP) period and it is not clear whether these induced changes will resolve over a longer period of time (i.e. in the upcoming months/years after delivery).

Understanding the cardiac adaptation during pregnancy and the reversal process in the postpartum period, as well as the factors that influence this these processes, may provide us not only insight in this mechanism, but may help us in identifying factors that may be target points for modification.

DETAILED DESCRIPTION:
The main goal of this study is to determine whether the presence of placental acute atherosis after pre-eclamptic pregnancies compared to normotensive pregnancies is related to the future development of subclinical atherosclerosis in the coronary arteries.

This information can be used to improve our prediction of which women have an increased risk of future cardiovascular disease and which women do not. This will allow us to better inform our postpartum population of the potential future risks of cardiovascular disease and could allow the timely implementation of primary prevention strategies. The investigators would also like to determine which blood biomarkers can also predict cardiovascular disease at an earlier stage as well as determining which of these biomarkers are present in hypertensive pregnancies.

This study is a longitudinal cohort study including women with pre-eclamptic pregnancies and normotensive pregnancies. Cases consist of women with preeclampsia (PE) and/or HELLP syndrome in the current pregnancy (early and late PE, with or without intra uterine growth restriction (IUGR)), whereas controls are women with an uncomplicated pregnancy.

The placenta is collected after the delivery and undergoes histopathological analyses. There are two follow up periods whereby one group of women is followed up 6 to 36 months postpartum and another group is followed up 10 to 20 years postpartum. At the follow up (6 to 36 months or 10 to 20 years), women attend for a series of measurements including CT angiography, transthoracic echocardiography, Flow medicated dilatation (FMD) and carotid intima media thickness (IMT) measurement. The visit will last approximately 5 hours in the Maastricht University Medical Centre (MUMC+). The only invasive procedure is a venepuncture where 75 ml blood will be extracted. The only unfavourable side effect can be a small hematoma (rare). Clinically, participants will be advised based on their risk profile following standard "cardiovascular (CV) risk management". Glycocalyx measurements and a FibroScan may be performed. Experience shows that this investigation is not experienced as uncomfortable. Also, 3 liters of exhaled air may be collected for volatile organic compound (VOCs) analysis. All measurements will be performed or supervised by an experienced researcher. These investigations are already approved previously in other Medical Ethics Committee (METC) applications (CMO-nr: 2008/226; 2009/004; 10-2-066). The other measurements (questionnaires, blood pressure (BP), weight measurement, urine collection, glycocalyx measurement, FibroScan and exhaled air collection) do not cause any discomfort for the patient aside from the time that it takes. On the other hand, potential health improvement and early detection of CV risk profiles and initiation of already existing effective prevention strategies that improve lifestyle are important benefits.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Controls: Women with an uncomplicated pregnancy at the moment of inclusion (i.e no foetal or maternal placental complications, such as pregnancy induced hypertension, preeclampsia or HELLP-syndrome, or small for gestational birth infancies)
* Cases: Women diagnosed with a preeclamptic pregnancy at the moment of inclusion

Exclusion Criteria:

• Women who do not want to be informed about the results of the tests, or women who do not want their general practitioner and specialist(s) to be informed about the test results

* Allergy or intolerance to glyceryl trinitrate, betablockers or iodinated contrast media.
* Controls: Pre-existing chronic hypertension treated with antihypertensive medication or autoimmune disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of pregnant women who either develop pre-eclampsia or have a normotensive pregnancy. For the shorter follow up period, participants are recruited from the (labour) ward and from the outpatient clinic in MUMC+. Participants are also recruited externally from other hospitals if they contact us with an interest in this study.
  For the longer follow up period, case participants took part in an earlier study and agreed to be contacted for future studies. These participants were recruited through a letter with information about the study. Control participants were recruited when they contacted us with interest in this study.
Sampling Method: Probability Sample
Enrollment: 226 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between placental acute atherosis and subclinical coronary atherosclerosis at 1 year postpartum | 1 year
  Acute atherosis will be defined as the presence of subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as either present or absent.
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of acute atherosis will be compared with each of the subcategories of subclinical coronary atherosclerosis for the pre-eclamptic and normotensive groups at 1 year postpartum.
Relationship between placental acute atherosis and subclinical coronary atherosclerosis at 15 years postpartum | 15 years
  Acute atherosis will be defined as the presence of subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as either present or absent.
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of acute atherosis will be compared with each of the subcategories of subclinical coronary atherosclerosis for the pre-eclamptic and normotensive groups at 15 years postpartum.
Relationship between decidual vasculopathy and subclinical coronary atherosclerosis at 1 year postpartum | 1 year
  Decidual vasculopathy will be defined as the presence of subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. It will be measured as either present or absent.
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of decidual vasculopathy will be compared with each of the subcategories of subclinical coronary atherosclerosis for the pre-eclamptic and normotensive groups at 1 year postpartum.
Relationship between placental decidual vasculopathy and subclinical coronary atherosclerosis at 15 years postpartum | 15 years
  Decidual vasculopathy will be defined as the presence of subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. It will be measured as either present or absent.
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of decidual vasculopathy will be compared with each of the subcategories of subclinical coronary atherosclerosis for the pre-eclamptic and normotensive groups at 15 years postpartum.

SECONDARY OUTCOMES:
Relationship between placental acute atherosis and clinical coronary atherosclerosis at 1 year postpartum | 1 year
  Acute atherosis will be defined as subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as present or absent.
  Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Calcification score of their coronary arteries is based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 hounsfield units (HU), multiplying the area of calcium by a factor related to maximum plaque attenuation.
  The agatston score ranges from 0 and has no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk of coronary events, >400 = high risk of coronary events.
  The incidence of acute atherosis will be compared with the average agatston score for the pre-eclamptic and normotensive groups at 1 year postpartum.
Relationship between placental acute atherosis and clinical coronary atherosclerosis at 15 years postpartum | 15 years
  Acute atherosis will be defined as subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as present or absent.
  Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Calcification score of their coronary arteries is based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 HU, multiplying the area of calcium by a factor related to maximum plaque attenuation.
  The agatston score ranges from 0 and has no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk of coronary events, >400 = high risk of coronary events.
  The incidence of acute atherosis will be compared with the average agatston score for the pre-eclamptic and normotensive groups at 15 years postpartum.
Relationship between placental decidual vasculopathy and clinical coronary atherosclerosis at 1 year postpartum | 1 year
  Decidual vasculopathy defined as subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. (Present or absent) Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Calcification score of their coronary arteries is based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 HU, multiplying the area of calcium by a factor related to maximum plaque attenuation.
  Range 0 to no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk, >400 = high risk.
  The incidence of decidual vasculopathy compared with average agatston score for the pre-eclamptic and normotensive groups at 1 year postpartum.
Relationship between placental decidual vasculopathy and clinical coronary atherosclerosis at 15 years postpartum | 15 years
  Decidual vasculopathy defined as subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. (Present or absent) Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Calcification score of their coronary arteries based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 HU, multiplying the area of calcium by a factor related to maximum plaque attenuation.
  Range 0 to no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk, >400 = high risk.
  The incidence of decidual vasculopathy compared with average agatston score for the pre-eclamptic and normotensive groups at 15 years postpartum.
Incidence of placental acute atherosis at 1 year postpartum | 1 year
  Acute atherosis will be defined as the presence of subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as either present or absent.
  The incidence of acute atherosis will be compared for the pre-eclamptic and normotensive groups at 1 year postpartum.
Incidence of placental acute atherosis at 15 years postpartum | 15 years
  Acute atherosis will be defined as the presence of subendothelial lipid-filled foam cells on placental histopathological analysis. It will be measured as either present or absent.
  The incidence of acute atherosis will be compared for the pre-eclamptic and normotensive groups at 15 years postpartum.
Incidence of placental decidual vasculopathy at 1 year postpartum | 1 year
  Decidual vasculopathy will be defined as the presence of subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. It will be measured as either present or absent.
  The incidence of decidual vasculopathy will be compared for the pre-eclamptic and normotensive groups at 1 year postpartum.
Incidence of placental decidual vasculopathy at 15 years postpartum | 15 years
  Decidual vasculopathy will be defined as the presence of subendothelial lipid-filled foam cells, fibrinoid necrosis, mural hypertrophy, chronic perivasculitis, absence of spiral artery remodelling and/or persistence of intramural endovascular trophoblast in the third trimester on placental histopathological analysis. It will be measured as either present or absent.
  The incidence of decidual vasculopathy will be compared for the pre-eclamptic and normotensive groups at 15 years postpartum.
Incidence of subclinical coronary atherosclerosis at 1 year postpartum | 1 year
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of each of the subcategories of subclinical coronary atherosclerosis will be compared for the pre-eclamptic and normotensive groups at 1 year postpartum.
Incidence of subclinical coronary atherosclerosis at 15 years postpartum | 15 years
  Subclinical coronary atherosclerosis will be measured using CT contrast angiography. This will be measured visually and split into the following categories: any atherosclerosis, wall irregularities, soft plaque and calcified plaque/stenosis.
  The incidence of each of the subcategories of subclinical coronary atherosclerosis will be compared for the pre-eclamptic and normotensive groups at 15 years postpartum.
Incidence of clinical coronary atherosclerosis at 1 year postpartum | 1 year
  Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Each patient will receive a calcification score of their coronary arteries based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 HU, multiplying the area of calcium by a factor related to maximum plaque attenuation: 130-199 HU, factor 1; 200-299 HU, factor 2; 300-399 HU, factor 3; and ≥ 400 HU, factor 4.
  The agatston score ranges from 0 and has no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk of coronary events, >400 = high risk of coronary events.
  The average agatston score will be compared for the pre-eclamptic and normotensive groups at 1 year postpartum.
Incidence of clinical coronary atherosclerosis at 15 years postpartum | 15 years
  Clinical coronary atherosclerosis will be measured using CT contrast angiography and the agatston score. Each patient will receive a calcification score of their coronary arteries based on the calcification seen on the CT scan. This is a continuous scoring system.
  The Agatston method uses the weighted sum of lesions with a density above 130 HU, multiplying the area of calcium by a factor related to maximum plaque attenuation: 130-199 HU, factor 1; 200-299 HU, factor 2; 300-399 HU, factor 3; and ≥ 400 HU, factor 4.
  The agatston score ranges from 0 and has no upper maximum. 0 = absent, 1-100 = low risk of coronary events, 101-400 = medium risk of coronary events, >400 = high risk of coronary events.
  The average agatston score will be compared for the pre-eclamptic and normotensive groups at 15 years postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spaanderman, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center (MUMC+), Maastricht, Netherlands

REFERENCES:
- [Derived] Jansen G, Alers RJ, Janssen EB, Jorissen LM, Morina-Shijaku E, Severens-Rijvers C, van 't Hof A, van Drongelen J, Scholten RR, Al-Nasiry S, Stevens D, Ganzevoort W, Gordijn S, Cornette J, Mihl C, Kietelaer B, Ghossein-Doha C, Spaanderman ME. PlacEntal Acute atherosis RefLecting Subclinical systemic atherosclerosis in women up to 20 years after pre-eclampsia (PEARLS): research protocol for a cohort study. BMJ Open. 2025 May 24;15(5):e100542. doi: 10.1136/bmjopen-2025-100542. PMID 40413047